CLINICAL TRIAL: NCT04560361
Title: The Analgesic Effect of Electroacupuncture on Postherpetic Neuralgia: a Multicenter Randomized Controlled Trial
Brief Title: The Analgesic Effect of Electroacupuncture on Postherpetic Neuralgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Qianyan Liu, Principal Investigator, Nanjing University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020NL-103-02
Record Dates: First submitted 2020-09-01; First posted 2020-09-23 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Postherpetic Neuralgia
Keywords: Electroacupuncture; Postherpetic Neuralgia; Analgesic effect
MeSH Terms: conditions — Neuralgia, Postherpetic

STUDY DESIGN:
Intervention Model Description: Using the center stratification block randomization method, the center is used as the stratification factor, and subjects were randomly assigned to the electroacupuncture group and the sham electroacupuncture group at a ratio of 1:1. The central randomization system is used for randomization operations.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The randomization scheme is generated, validated and imported into the central randomization system by a statistician who do not participate in this trial by using R software. The central randomization system has set strict personnel permissions, and no one has right to view the randomization scheme except the highest-level system administrator. Patients and study investigators (i.e., outcome assessors, data recorders, data entry clerks and statistical analysts) will be blinded to the group assignment. Due to the nature of the intervention, acupuncturists will not be blinded to the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture group (Experimental): Choose the appropriate position according to the patient's herpes site, and routinely disinfect the skin. Paste the fixed insulating pad on the acupoint, and use a 0.30×40mm acupuncture needle to penetrate the skin 10mm obliquely through the fixed insulating gasket at Ashi point; According to the above operation, the SJ6 and GB34 point of the affected side are directly penetrated into the skin 15-20mm. The local Ashi point connects the two poles of the electroacupuncture device according to the first and last points of the long axis of the painful part, and the SJ6 and GB34 point on the affected side are connected to the poles of the electroacupuncture device. Electroacupuncture waveform is continuous wave, frequency is 2Hz, and current intensity is 1-5mA (causing slight tremor of the skin around the acupuncture point without pain). Continue the electroacupuncture treatment for 30 minutes.
  Interventions: Other: Electroacupuncture treatment
- Sham electroacupuncture group (Sham Comparator): Participants randomly assigned to the sham electroacupuncture (SA) group received sham electroacupuncture by using placebo blunt needles at the same acupoints. After disinfecting the skin and placing the sterile insulating adhesive pads on unilateral Zhigou, Yanglingquan and Ashi points, placebo blunt needles are inserted through the pads and reach the insulating adhesive layer, causing the participants to feel the needle resistance (a sensation of needle insertion). Other procedures, electrode placements, parameter of electroacupuncture apparatus and treatment settings are the same as in the EA group, but with no skin penetration or electricity output.
  Interventions: Other: Sham electroacupuncture treatment

INTERVENTIONS:
Other: Electroacupuncture treatment — Continue the electroacupuncture treatment as described above for 30 minutes.
  Arms: Electroacupuncture group
Other: Sham electroacupuncture treatment — Continue the sham electroacupuncture treatment as described above for 30 minutes.
  Arms: Sham electroacupuncture group

SUMMARY:
The investigators designed the multicenter randomized parallel controlled clinical trial of electroacupuncture on PHN which is rigorously designed and have an appropriate sample size, aiming to evaluate the efficacy and safety of electroacupuncture in pain relieving and pain removing in the treatment of patients with PHN.

DETAILED DESCRIPTION:
Postherpetic neuralgia(PHN) is the most common complication of herpes zoster, is a severe and intractable pain with a high incidence. Nearly 50% of PHN patients have experienced persistent pain for more than one year. Although it is not directly life-threatening, will lead to sleep disorders, even depression, seriously affecting the quality of life of patients. This project is a multi-center randomized controlled trial, which will recruit 448 patients with PHN in 7 hospitals, aiming to evaluate the analgesic effect and safety of electroacupuncture on postherpetic neuralgia, and provide evidence-based medical evidence for electroacupuncture treatment of PHN.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet the diagnostic criteria for postherpetic neuralgia (with a clear history of acute herpes zoster, and the duration of postherpetic pain exceeds 90 days)
* Aged 45 to 75 years old
* Patients who were diagnosed with moderate or above pain during the observation period (the daily pain score was continuously collected within 7 days during the observation period, and the average NRS-11 pain score was >=4)
* Subjects who did not participate in other ongoing clinical studies
* Sign informed consent and volunteer to participate in the study

Exclusion Criteria:

* Patients who are currently receiving or receiving more than one of the "permitted combinations" or any "prohibited combination and treatment" for PHN listed in the following part at least 14 days before screening, and are unwilling to undergo washout period, or patients with serious safety problems during washout period or observation period
* Patients who are expected to receive any new prescription drug or other treatment for PHN after the start of the trial
* Patients with serious uncontrolled medical conditions, such as cardiovascular, lung, liver, kidney, gastrointestinal tract, metabolism, endocrine, nervous system, respiratory system, urogenital system and other serious diseases, or systemic organ dysfunction, malignant tumor, hematologic disease such as bleeding tendency or coagulation dysfunction, serious mental illness such as depression or schizophrenia Symptoms, hepatitis B antigen or hepatitis C antibody positive known state or history of immune dysfunction, history of HIV infection, etc.
* Patients with severe pain unrelated to PHN, such as after surgery for clinical major diseases
* Patients with PHN who have received nerve intervention or other neurosurgical treatment, such as selective nerve damage, percutaneous radiofrequency thermocoagulation or pulsed nerve modulation technology, etc.
* Patients with some special types of herpes zoster, such as those with meninges, cornea, conjunctiva, ear involvement, visceral herpes zoster, generalized herpes zoster
* Patients with skin ulceration, new herpes, or skin infection
* Patients with cardiac pacemaker, metal allergy or severe fear of needle
* Patients who are unable to give full informed consent or cannot cooperate with pain scale assessment due to mental, mental, linguistic or behavioral disorders
* Patients who have poor compliance or are prone to fall off due to other reasons, such as the current residence is not in the city where the recruitment hospital is located, or the working environment changes frequently
* Pregnant and lactating women

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2022-08-23 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity (NRS-11) | Change from Baseline at 4 weeks after treatment
  11-point numeric rating scale (NRS-11): range from 0 (no pain) to 10 (worst possible pain), with 1-3 points representing mild pain, 4-6 points representing moderate pain, and 7-10 points representing severe pain. A reduction of ≥30% in NRS-11 scores from baseline were considered responders.

SECONDARY OUTCOMES:
Change in pain intensity (VAS) | Change from Baseline at 1 day, 3 days, 1 week, 2 weeks, 3 weeks and 4 weeks after treatment
  Visual analogue scale (VAS): a horizontal line without verbal descriptors or numbers at intermediate points (0=no pain, 10=worst imaginable pain)
Change in the interference of pain on sleep | Change from Baseline at 1 day, 3 days, 1 week, 2 weeks, 3 weeks and 4 weeks after treatment
  Verbal rating scale (VRS): 4 levels.
  1. Level 0: No pain.
  2. Level I (mild): Pain but tolerable, normal life, no interference with sleep.
  3. Level II (moderate): Pain is obvious, unbearable, requires analgesic medication, and sleep is disturbed.
  4. Level III: Severe pain, unbearable, analgesic medication, severe interference with sleep, accompanied by autonomic dysfunction or passive positions.
Change in mechanical pain threshold (MPT) | Change from Baseline at 1 day, 3 days, 1 week, 2 weeks, 3 weeks and 4 weeks after treatment
  Stimulated the most painful central part of PHN with a series of von Frey hairs (0.008-300 g).
Change in pain area of PHN (PAP) | Change from Baseline at 1 day, 3 days, 1 week, 2 weeks, 3 weeks and 4 weeks after treatment
  calculated by the researcher based on 45 body areas rating scale (BARS-45) which requires the use of height and weight of the patient.
Change in average number of pain episodes per day | Change from Baseline at 1 day, 3 days, 1 week, 2 weeks, 3 weeks and 4 weeks after treatment
  Painless: 0 times; Intermittent pain: 1-50 times (1-2, 3-5, 6-10, 11-50 optional); Persistent pain: >50 times.
Change in average duration of each pain episode (ADEPE) | Change from Baseline at 1 day, 3 days, 1 week, 2 weeks, 3 weeks and 4 weeks after treatment
  Duration ranges from 0 minutes (no pain) to 24 hours (persistent pain).
Change in the nature and intensity of pain | Change from Baseline at 4 weeks after treatment
  short form of McGill pain questionnaire 2 (SF-MPQ-2): includes 22 items.
Change in degree of pain and its impact on work life, interpersonal relationships and sleep | Change from Baseline at 4 weeks after treatment
  Zoster brief pain inventory (ZBPI)
Change in depression, anxiety and positive outlook scale (DAPOS) | Change from Baseline at 4 weeks after treatment
  11 items, combines depression (5 items), anxiety (3 items) and positive outlook (3 items).
Change in overall impression of PHN | 4 weeks
  Patient global impression of change (PGIC): Participants were asked to describe their overall impression of change of their condition/pain by answering the following question: "Compared to your pain at admission to the project, how much has it changed?" (categories: much improved = 1, mildly improved = 2, unchanged = 3, mildly worsened = 4, much worsened = 5).

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Sun, Study Director — Jiangsu Province Hospital of Traditional Chinese Medicine; Wenping Yao, Principal Investigator — Lianyungang Hospital of Traditional Chinese Medicine; Yongtao Liu, Principal Investigator — Huai'an Hospital of Traditional Chinese Medicine; Juanjuan Shi, Principal Investigator — Affiliated Hospital of Nanjing University of Chinese Medicine; Hua Feng, Principal Investigator — Wuxi Hospital of Traditional Chinese Medicine; Chunxia Lu, Principal Investigator — Nantong Hospital of Traditional Chinese Medicine; Yanfang Liu, Principal Investigator — Shuyang Hospital of Traditional Chinese Medicine
Locations (7):
- China (7):
  - Huai'an Hospital of Traditional Chinese Medicine, Huai'an, Jiangsu
  - Lianyungang Hospital of Traditional Chinese Medicine, Lianyungang, Jiangsu
  - Nanjing Hospital of Chinese Medicine Affiliated to Nanjing University of Chinese Medicine, Nanjing, Jiangsu
  - Jiangsu Province Hospital of Chinese Medicine, Nanjing, Jiangsu
  - Nantong Hospital of Traditional Chinese Medicine, Nantong, Jiangsu
  - Shuyang Hospital of Traditional Chinese Medicine, Suqian, Jiangsu
  - Wuxi Hospital of Traditional Chinese Medicine, Wuxi, Jiangsu

IPD SHARING:
Plan to Share IPD: Yes
Case Report Form, Electronic Data Capture(EDC)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within six months after the trial complete
Access Criteria: Use the EDC system of the Science and Technology Department of Jiangsu Provincial Hospital of Chinese Medicine to disclose the original data
URL: http://jshtcm.ecrfdata.com/edc/inx/jshtcm

REFERENCES:
- [Background] van Hecke O, Austin SK, Khan RA, Smith BH, Torrance N. Neuropathic pain in the general population: a systematic review of epidemiological studies. Pain. 2014 Apr;155(4):654-662. doi: 10.1016/j.pain.2013.11.013. Epub 2013 Nov 26. PMID 24291734
- [Background] Kawai K, Gebremeskel BG, Acosta CJ. Systematic review of incidence and complications of herpes zoster: towards a global perspective. BMJ Open. 2014 Jun 10;4(6):e004833. doi: 10.1136/bmjopen-2014-004833. PMID 24916088
- [Background] Wang L, Qiu L, Zheng X, Ouyang J, Zhang M, He L, Zeng S, Liu B, Peng J. Effectiveness of electroacupuncture at Jiaji acupoints (EX-B2), plus moxibustion and intermediate on postherpetic neuralgia: a randomized controlled trial. J Tradit Chin Med. 2020 Feb;40(1):121-127. PMID 32227773
- [Background] Wu CH, Lv ZT, Zhao Y, Gao Y, Li JQ, Gao F, Meng XF, Tian B, Shi J, Pan HL, Li M. Electroacupuncture improves thermal and mechanical sensitivities in a rat model of postherpetic neuralgia. Mol Pain. 2013 Apr 3;9:18. doi: 10.1186/1744-8069-9-18. PMID 23551937
- [Background] Pei W, Zeng J, Lu L, Lin G, Ruan J. Is acupuncture an effective postherpetic neuralgia treatment? A systematic review and meta-analysis. J Pain Res. 2019 Jul 16;12:2155-2165. doi: 10.2147/JPR.S199950. eCollection 2019. PMID 31410050
- [Background] Werner RN, Nikkels AF, Marinovic B, Schafer M, Czarnecka-Operacz M, Agius AM, Bata-Csorgo Z, Breuer J, Girolomoni G, Gross GE, Langan S, Lapid-Gortzak R, Lesser TH, Pleyer U, Sellner J, Verjans GM, Wutzler P, Dressler C, Erdmann R, Rosumeck S, Nast A. European consensus-based (S2k) Guideline on the Management of Herpes Zoster - guided by the European Dermatology Forum (EDF) in cooperation with the European Academy of Dermatology and Venereology (EADV), Part 1: Diagnosis. J Eur Acad Dermatol Venereol. 2017 Jan;31(1):9-19. doi: 10.1111/jdv.13995. Epub 2016 Nov 2. PMID 27804172
- [Background] Hjermstad MJ, Fayers PM, Haugen DF, Caraceni A, Hanks GW, Loge JH, Fainsinger R, Aass N, Kaasa S; European Palliative Care Research Collaborative (EPCRC). Studies comparing Numerical Rating Scales, Verbal Rating Scales, and Visual Analogue Scales for assessment of pain intensity in adults: a systematic literature review. J Pain Symptom Manage. 2011 Jun;41(6):1073-93. doi: 10.1016/j.jpainsymman.2010.08.016. PMID 21621130
- [Derived] Liu Q, Wu X, Guo J, Gao J, Liu B, Wang Y, Xia M, Pei L, Sun J. Analgesic Effect of Electroacupuncture on Postherpetic Neuralgia: A Trial Protocol for a Multicenter Randomized Controlled Trial. Pain Ther. 2021 Dec;10(2):1755-1771. doi: 10.1007/s40122-021-00283-8. Epub 2021 Jul 12. PMID 34254233

DOCUMENTS (1):
  • Study Protocol (2021-04-15): https://cdn.clinicaltrials.gov/large-docs/61/NCT04560361/Prot_000.pdf